CLINICAL TRIAL: NCT06156735
Title: The Effect of Music Therapy on Cognition in Neurorehabilitation - A Feasibility Randomized Controlled Trial
Brief Title: Music Therapy on Cognition in Neurorehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Record Dates: First submitted 2023-08-02; First posted 2023-12-05 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Dementia; Stroke; Traumatic Brain Injury
Keywords: Music therapy; Active; Passive; neurorehabilitation needs; Cognition
MeSH Terms: conditions — Dementia; Stroke; Brain Injuries, Traumatic; Motor Activity

STUDY DESIGN:
Intervention Model Description: participant will receive one passive music therapy session consisting of relaxation to music, one active music therapy session consisting of instrument-playing, and one control condition.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Passive Music Therapy (P) (Experimental): The therapist read a standardized relaxation script in the research participant's selected preferred language while improvising on the keyboard. The script was inclusive of deep breathing and imagining a positive image. The research participants were asked to close his or her eyes while relaxing and imagining. The entire intervention lasted approximately 15 minutes. The research participants were allowed to request to stop the intervention at any time
  Interventions: Other: Passive Music Therapy (P)
- Active Music Therapy (A) (Experimental): The research participants were given a standardized assortment of percussion instruments to choose from. The therapist provided instructions of playing instruments along with the therapist. The research participant was allowed to change his or her instrument at any time and was advised to sing along with the therapist. Based on the research participant's age, the therapist selected the songs to sing and accompany on either the guitar or the keyboard. The duration of the intervention was approximately 15 minutes, which allowed about five to six songs to be sung. The research participants were allowed to request to repeat or skip any of the songs at any time.
  Interventions: Other: Active Music Therapy (A)
- Standard Care Control Condition (C) (Active Comparator): The control condition involved mundane activities such as chatting, resting, or reading magazines, with the MT, in the treatment room.
  Interventions: Other: Standard Care Control Condition (C)

INTERVENTIONS:
Other: Passive Music Therapy (P) — Music Therapy Intervention
  Arms: Passive Music Therapy (P)
Other: Active Music Therapy (A) — Music Therapy Intervention
  Arms: Active Music Therapy (A)
Other: Standard Care Control Condition (C) — Without any intervention
  Arms: Standard Care Control Condition (C)

SUMMARY:
Music therapy has received more attention with its surging application in neuro-rehabilitation overseas. Given the dearth of music therapy and cognitive rehabilitation research conducted in Malaysia, this pilot study intended to investigate the effect of active and passive music therapy interventions versus the standard care condition in cognition among adults with neuro-rehabilitation needs.

DETAILED DESCRIPTION:
Music therapy has received more attention with its surging application in neuro-rehabilitation overseas. Given the dearth of music therapy and cognitive rehabilitation research conducted in Malaysia, this pilot study intended to investigate the effect of active and passive music therapy interventions versus the standard care condition in cognition among adults with neuro-rehabilitation needs.

Thirty subjects participated in this study. Each participant received one session of each of the following: active music therapy intervention, passive music therapy intervention, and standard card. Mini-Cog tests were conducted before and after each session and the scores were collected for data analysis. Throughout the study, observations ensured the troubleshooting of any potential flaws for future recommendations.

ELIGIBILITY:
Inclusion Criteria:

* NeuroRehabilitation Needs

Exclusion Criteria:

* obtain a score of above 22 or below 10 on the MMSE
* have documented current/active episodes of hallucinations and/or delusions
* have documented hearing impairments with or without hearing aid(s)
* have language barrier, i.e. do not speak or understand English, Mandarin or Malay

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Mini-Cog™ test | 1 year
  The Friedman test was conducted to determine whether Mini-Cog test scores differ from P, A, and C. A score of 0-2 suggests a higher likelihood of significant cognitive impairment, while a score of 3-5 indicates a lower likelihood of dementia but does not exclude mild impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- SOSCO Rehabilitation Centre, Malacca, Malacca, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT06156735/Prot_SAP_002.pdf
  • Informed Consent Form (2025-04-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT06156735/ICF_003.pdf